CLINICAL TRIAL: NCT04806191
Title: Making Shoulder Pain Simple in General Practice-implementing an Evidenced Based Guideline for Shoulder Pain, a Hybrid Design Cluster Randomised Study
Brief Title: Simple and Evidence-based Examination and Treatment of Shoulder Pain in General Practice
Acronym: EASIER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: Helse Fonna (Other)
Responsible Party: Principal Investigator, Niels Gunnar JUEL, MD. PhD, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019/104
Record Dates: First submitted 2021-03-03; First posted 2021-03-19 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Pain; Frozen Shoulder; Rotator Cuff Tendinosis; Myalgia; Rotator Cuff Impingement Syndrome; Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: General practice; Implementation; Guideline
MeSH Terms: conditions — Shoulder Pain; Bursitis; Rotator Cuff Injuries; Myalgia; Shoulder Impingement Syndrome; Rupture | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded for treatment allocation. Randomization will be done after recruitment of GPs. GPs and study coordinators and outcome evaluators will be blinded to the allocation sequence with only the allocation of the next GP surgery being revealed by randomization list holder approximately 6 weeks before each intervention implementation point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be assessed by GPs who have attended an outreach workshop and trained at using an evidence based strategy for shoulder examination and treatment. GPs will have access to a decision support tool and patients is offered a tailored information package for self management.
  Interventions: Other: Evidence based treatment strategy; Other: Targeted patient information package
- Treatment as usual (TAU) (Active Comparator): The participants enrolled in the control period will receive treatment as offered in general practice.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Other: Evidence based treatment strategy — Evidence-based clinical examination and treatment plan
  Arms: Intervention
Other: Targeted patient information package — GPs will in cooperation with the patients tailor a information package targeted to the patients needs regarding their clinical shoulder diagnosis and individual implications and needs (Pain, sleep, exercises etc.).
  Arms: Intervention
Other: Treatment as usual (TAU) — Usual care as provided by the GP
  Arms: Treatment as usual (TAU)

SUMMARY:
Previous research suggests that general practitioners find handling patients with shoulder pain difficult and that the current care for shoulder pain is not in line with the best available evidence (1).This project aims to assess the effectiveness, costs and implementation of an evidence-based guideline for shoulder pain in general practice.

DETAILED DESCRIPTION:
A simplified and evidence-based algorithm for examination and treatment of patients with shoulder pain will be developed and implemented in general practice. The purpose is to improve quality of care and provide GPs with a simplified and efficient tool to handle patients with common shoulder- related pain. The study is a stepped-wedge, cluster-randomized trial with a hybrid design including a effectiveness, cost and implementation assessment of a guideline-based intervention in clinical practice (2). General practitioners in Norway will be recruited and the GP offices will be randomized to the time of crossover from current treatment as usual (TAU) to the implementation of the intervention. The intervention is a tailored strategy that includes workshops for general practitioners covering information and access to a decision support tool, an education program where the general practitioner learn an evidence-based approach to shoulder pain and access to patient information materials. Outcomes will be measured at patient and GP levels, using self-report questionnaires, focus group interviews and register based data.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the shoulder region
* Above 18 years

Exclusion Criteria:

* Unable to fill in self-report questionnaires or do not understand Norwegian
* Acute injury with clinical suspicion of fracture, luxation of shoulder joints or large tendon ruptures
* Clinical suspicion of referred pain to the shoulder area from other organs
* Signs of inflammatory joint disease
* Suspicion of malignant disease
* Symptoms and signs of cervical radiculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | Change from 0 to 12 weeks
  13 item patient reported questionnaire on shoulder pain and disability. (0 = no pain or shoulder disability, 100 = worst pain and disability).

SECONDARY OUTCOMES:
the EuroQol quality of life measure (EQ5D-5L) | Change from 0 weeks to 52 weeks
  Health related quality of life ((0 (death) - 1.0 (perfect health))
Patient reported quality of care index (treatment according to the guideline intervention) | 0 week (after 1. visit to general practitioner)
  Patient reported content of treatment measured on six items according to treatment prescribed by the GP measured on 5-item Likert scales. Sum score above 18 points regarded as consultation of high quality according to guideline intervention.
Global patient perceived effect of treatment outcome (GPE) | Measured at 6,12 and 52 weeks. Primary analysis of interest is at 12 weeks.
  1 item (7-point) ( 0 = worse than ever, 7 =I have become completely well)

OTHER OUTCOMES:
Brief illness perception questionnaire (BIPQ) | Measured at 0, 6, 12, 52 weeks, Primary time point of interest is 12 weeks and analysing changescore from 0 to 12 weeks.
  Illness perception 0-80 where a higher score reflects a more threatening view of the illness
Pain self-efficacy questionnaire (PSEQ) | Measured at 0, 6, 12, 52 weeks, primary time point of interest is 12 weeks analysing change score from 0 to 12 weeks.
  Self efficacy for pain 0-60 where higher score reflects higher self efficacy for pain.
Work disability patient reported | Measured at 0, 6, 12, 52 weeks
  Sick leave reported as whole days away from work
Örebro Musculoskeletal Pain Screening Questionnaire (Short) | Measured at 0 weeks
  Psychosocial, prognostic factors for musculoskeletal pain. The total score will range between 1 and 100, with a score >50 indicating higher estimated risk for future work disability
Pateint reported frequency of therapy due to shoulder pain in primary and secondary health care | Measured at 0, 6, 12, 52 weeks
  Reported number of consultations by GPs, specialists (orthopeds, rheumatologists, physiatrists or neurologists), physiotherapists, chiropractists and alternative therapists, injections and surgery.
Patient reported frequency of use of supplemental investigations in primary and secondary health care. | Measured at 0, 6, 12, 52 weeks
  Number of investigations; blood tests and radiology (Projectional radiograph, CT, MRI)
Patient reported direct economical expences due to shoulder pain | Measured at 0, 6, 12, 52 weeks
  Patient reported use of medication reported as type of medication and frequency last week
Patient reported indirect economical expences due to shoulder pain; travel distance to therapy | Measured at 0, 6, 12, 52 weeks
  Patient reported travel distance to therapy measured in km
Patient reported indirect economical expences due to shoulder pain; time away for therapy measured in hours | Measured at 0, 6, 12, 52 weeks
  Patient reported time away for therapy measured in hours
Patient reported indirect economical expences due to shoulder pain; time away for work measured in hours. | Measured at 0, 6, 12, 52 weeks
  Patient reported time away from work measured in hours
Patient reported indirect economical expences due to shoulder pain; production loss. | Measured at 0, 6, 12, 52 weeks
  Patient reported production loss measured as patient estimated per cent production loss due to shoulder pain. A higher number means a higher loss of production.
Work disability from the Norwegian Labour and Welfare Administration registry | Measured at 52 weeks
  Registry data
Global patient perceived satisfaction with treatment | Measured at 6, 12, 52 weeks
  1 item (5-point Likert scale); 0=dissatisfied, 5=very satisfied
Patient experience questionnaire (PEQ) | Measured at 0 weeks
  4 subscales (communication, emotions, outcome, barriers) with 4 items measured on 4 or 7 point Likert scales. A high score represents a good communication experience, positive emotions, positive consultation outcome, no communication barriers.
Patient Shoulder Outcome Expectancies | Measured at 0 week, 12 weeks
  1 item measured on a 7-point Likert scale. A higher score indicate higher patient perceived outcome expectancy.
Patient interview (qualitative) | Measured at 52 weeks
  Qualitative interview with selected patients, feasibility/ barriers and facilitators
Implementation process assesment tool (IPAT) | Measured at 2 weeks, 12 weeks
  Measurement of the implementation process from the perspective of the GPs
GPs self-efficacy for handling patients with shoulder pain according to guideline care | Measured at 0 week, 2 weeks,12 weeks
  9 items measured on 6-point Likert scales analysing change in individual items and sum score before and 12 weeks after educational outreach. A higher score indicates higher self-efficacy
GPs global perceived satisfaction with workshop (GP) | Measured at 0 weeks
  10 item measured on 5-point Likert scales concerning satisfaction with the different topics and content of the work shop.We will analyze individual items. A higher score indicate higher satisfaction.
GPs global perceived satisfaction, benefit, usability and frequency of use of the intervention (GP) | Measured at 12 weeks
  4 item measured on 5-point Likert scales. We will analyze individual items. A higher score indicate higher satisfaction, benefit, usability and frequency of use of the intervention.
GPs use of the intervention in daily practice; degree of simplifying shoulder evaluation and treatment, recommending exercises, information and patient involvement (GP) | Measured at 12 weeks
  4 items measured on 7-point Likert scales. We will analyze individual items. A higher score indicate higher degree of use in daily practice and a higher degree of simplifying shoulder evaluation and treatment, recommending exercises, information and patient involvement.
GP focus groups | Measured at 52 weeks
  Qualitative interview with selected GPs, feasibility/ barriers and facilitators

CONTACTS AND LOCATIONS:
Overall Officials: Niels G Juel, MD, PhD, Principal Investigator — Department of General practice, University of Oslo
Locations (2):
- Norway (2):
  - Department of Research and innovation, Helse Fonna, Norway, Haugesund, Vestland
  - Department of General Practice, University of Oslo, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Artus M, van der Windt DA, Afolabi EK, Buchbinder R, Chesterton LS, Hall A, Roddy E, Foster NE. Management of shoulder pain by UK general practitioners (GPs): a national survey. BMJ Open. 2017 Jun 21;7(6):e015711. doi: 10.1136/bmjopen-2016-015711. PMID 28637737
- [Derived] Ekeberg OM, Pedersen SJ, Natvig B, Brox JI, Biringer EK, Endresen Reme S, Engebretsen KB, Joranger P, Mdala I, Juel NG. Making shoulder pain simple in general practice: implementing an evidence-based guideline for shoulder pain, protocol for a hybrid design stepped-wedge cluster randomised study (EASIER study). BMJ Open. 2022 Jan 7;12(1):e051656. doi: 10.1136/bmjopen-2021-051656. PMID 34996788